CLINICAL TRIAL: NCT04882488
Title: Correlation of FFR and iFR With Cardiac PET Perfusion (at Rest and Under Adenosine) in the Evaluation of Intermediate Coronary Stenoses in Patients With Severe Aortic Valve Stenosis
Brief Title: Correlation of FFR and iFR With Cardiac PET Perfusion in Patients With Severe Aortic Valve Stenosis
Acronym: TAVI PET
Status: Recruiting | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: HDZ-KA_020_TR
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Aortic Valve Stenosis; Coronary Artery Disease
Keywords: Aortic valve stenosis; PET-CT; coronary artery disease; FFR
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — NT pro BNP,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aortic valve stenosis (AS) affects 2-7% of persons > 65 years, symptoms include: angina and dyspnea, dizziness and syncope. Coincidence of coronary artery disease (CAD), also presenting with angina and dyspnea, in patients with AS between 40 - 65% . Angina in AS caused by significant reduction of coronary flow reserve (CFR). CFR is the ratio of maximal flow increase in the coronary vessel bed during maximal hyperaemia (medically or exercise induced). FFR (fractional flow reserve) use in patients with AS potentially invalid due to dysfunctional CFR leading to potential undertreatment of CAD in these patients.CFR disturbance in AS mainly due to myocardial overload causing concentric hypertrophy, increased oxygen consumption and neurohormonal activation leading to increased vascular resistance. Current studies are investigating the validity of FFR and iFR in AS patients. Recent data demonstrate very good correlation between FFR and iFR derived values to PET myocardial perfusion imaging values in patients with no evidence of AS. Our study aims to investigate the diagnostic performance of FFR and iFR in intermediate-grade coronary stenosis in patients with severe aortic valve disease and correlate FFR- and iFR derived values with those extracted from PET-perfusion Imaging.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe aortic Stenosis eligible for transcatheter aortic stenosis
* left ventricular ejection fraction > 55%
* no intolerance of Adenosin
* no history of bradycardia, atrioventricular Blockade
* intermediate coronary Stenosis with FFR> 0.8
* Age >65

Exclusion Criteria:

* intolerance of Adenosin
* left ventricular ejection fraction < 55%

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with severe aortic Stenosis eligible for transcatheter aortic Valve Implantation (TAVI) with concurring coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of PET-CT Prior to TAVI and 3 months after TAVI procedure | 3 months
  Evaluation of FFR-negative intermediary coronary stenoses in Patients with severe Aortic Stenosis Prior and 3 months following TAVI

SECONDARY OUTCOMES:
Clinical Evaluation Prior to and following TAVI | 3 months
  Angina prevalence in patients with intermediate coronary Stenosis Prior to and 3 months following TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Rudolph, MD, Principal Investigator — Consultant physician
Locations (1):
- Herz- und Diabeteszentrum, NRW, Bad Oeynhausen, North Rhine-Westphalia, Germany